CLINICAL TRIAL: NCT05726630
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study of the Efficacy and Safety of Divozilimab in Patients With Systemic Scleroderma
Brief Title: Clinical Study of Divozilimab in Patients With Systemic Scleroderma
Acronym: LIBERIUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-132-5
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-11

CONDITIONS: Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Divozilimab (Experimental)
  Interventions: Drug: Divozilimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Divozilimab — anti CD20 monoclonal antibody
  Arms: Divozilimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled clinical study of the efficacy and safety of divozilimab in patients with systemic scleroderma.The study will enroll adult patients of both sexes diagnosed with active systemic scleroderma according to the ACR/EULAR 2013 criteria with a modified Rodnan skin score (mRSS) of 10 to 20. In patients having signs of ILD, the Forced Vital Capacity (FVC) should be at least 40 % of the due value. Subjects will be randomized to divozilimab or placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "systemic scleroderma" in accordance with the ACR/EULAR 2013 classification.
* Modified Rodnan skin score (mRSS) from 10 to 20.
* FVC ≥ 40 % of the due value.

Exclusion Criteria:

* Induced scleroderma.
* Silicone implants/protheses.
* Digital ulcers with signs of infection or indications for any amputation.
* Blood biochemistry or hematological abnormalities at screening.
* FEV1/FVC < 0.7 and FEV1< 50 % at screening.
* History of threatment with anti-CD20 monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in the modified Rodnan Skin Score (mRSS) from baseline | week 24
  The modified Rodnan Skin Score (mRSS) describes the thickness of skin in 17 anatomic areas rated from 0 to 3, where 3 indicates the most severe thickening.

SECONDARY OUTCOMES:
Change in the modified Rodnan Skin Score (mRSS) from baseline | week 48
  The modified Rodnan Skin Score (mRSS) describes the thickness of skin in 17 anatomic areas rated from 0 to 3, where 3 indicates the most severe thickening.
Change in the FVC (forced vital capacity) from baseline | week 48
  Forced vital capacity is the amount of air that can be forcibly exhaled after the deepest possible breath.
Change in Health Assessment Questionnaire Disability Index (HAQ-DI) score from baseline | week 48
  Change in Health Assessment Questionnaire Disability Index (HAQ-DI) describes the patient's self-assessed degree of disability. HAQ-DI comprises 8 categories of questions rated from 0 to 3, where 3 indicates the worst degree of disability.

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - Clinical Rheumatology Hospital №25, Saint Petersburg
  - North-Western state Medical University named after I.I. Mechnikov, Saint Petersburg